CLINICAL TRIAL: NCT03214744
Title: Rapid Versus Slow Entral Feeding Advancements on Clinical Outcomes of Preterm Infants
Acronym: pretermfood
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amany Makrm Riad, Rapid Versus Slow Entral Feeding Advancements on Clinical Outcomes of Preterm Infants, Assiut University
Other Study IDs: 17100036
Record Dates: First submitted 2017-07-09; First posted 2017-07-12 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Preterm Infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rapid Versus Slow Entral Feeding Advancements on Clinical Outcomes of Preterm Infants

DETAILED DESCRIPTION:
Rapid feeding advancement achieves full enteral volume of feedings earlier than the slower advancement.They received significantly fewer days of parenteral nutrition, exhibited a shorter time to regain birth weight and shorter duration of hospital stay. The incidence of NEC and the number of episodes of feeding intolerance were not significantly different between rapid and slow advancement. while the incidence of culture-proven late onset sepsis was significantly less in infants receiving a rapid feeding advancement

ELIGIBILITY:
Inclusion Criteria:

- All preterm neonates admitted to NICU with gestational age less than 36 weeks, and haemodynamically stable

Exclusion Criteria:

* gastrointestinal tract anomalies,
* haemodynamically unstable infants,
* gestatinal age equal or more than 36 weeks,
* preterms who develop NEC,
* preterms on mechanical ventilation.

Ages: 1 Week to 15 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates (<36 weeks)
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
effect of entral feeding on preterm | six months
  -Length of hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: John J Smith, Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- Assiut university, Asyut, Egypt

REFERENCES:
- [Background] Pike K, Brocklehurst P, Jones D, Kenyon S, Salt A, Taylor D, Marlow N. Outcomes at 7 years for babies who developed neonatal necrotising enterocolitis: the ORACLE Children Study. Arch Dis Child Fetal Neonatal Ed. 2012 Sep;97(5):F318-22. doi: 10.1136/fetalneonatal-2011-300244. PMID 22933088